CLINICAL TRIAL: NCT06505434
Title: A Dynamic Study of Pupil Diameter After Artificial Lens Implantation in Patients With High Myopia
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: QX-2023-A-011
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cataract
Keywords: cataract; high myopia
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low myopia group: A low myopia group (0D to -6.0D)
  Interventions: Procedure: Cataract surgery
- high myopia group: B high myopia group (-6.0 to -12.0D)
  Interventions: Procedure: Cataract surgery
- ultra-high myopia group: C ultra-high myopia group (greater than -12.0D) group
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Phaco + IOL Implantation

SUMMARY:
Age-related cataract remains the leading cause of blindness in developing countries. And, with the aging of the population in these countries, the number of cataract patients will continue to grow. With accurate biological measurements and the implantation of appropriate IOLs, most cataract patients can achieve good distance vision after surgery. However, it should not be overlooked that the current global prevalence of myopia is over 28.3% and is expected to reach 49.8% by 2050, while the rate of high myopia will increase from the current 4.0% to 9.8%. The prevalence of cataracts is significantly higher in the highly myopic population than in the orthoptic population.

The pupil is an important factor to be evaluated during the selection of an artificial lens (Intraocular lens, IOL), especially a functional IOL. It has been shown that the diameter and sensitivity of the pupil in patients with high myopia are also significantly different from those in the orthopneic population, and that there is a correlation with the adjustment status and refractive error. The purpose of this study is to investigate the following: 1. Whether the change of refractive status before and after IOL implantation in highly myopic cataract patients will lead to the change of pupil physiological characteristics, and whether the modification of preoperative measurement parameters can expand the population of myopic patients who can be reasonably applied to the functional IOL and obtain a high degree of satisfaction from patients. 2. Pupil diameter under a single fixed light source is a rough assessment for the screening of the population for functional IOLs, and this study was conducted in a single fixed light source. In this study, we measured the maximum value of pupil diameter, minimum value of pupil diameter, and rate of change of pupil diameter under bright vision and dark vision, and analyzed the correlation between the above three parameters and visual quality to further optimize the objective index of pupil diameter for the screening of functional IOL applicants.

Objectives of the study

1. To observe the dynamic changes of pupil diameter and its visual quality before and after lens extraction combined with IOL implantation in myopic patients, and to analyze the correlation between the changes of pupil diameter and visual quality;
2. To explore the patterns of refractive error and pupil biometric changes in myopic patients before and after IOL implantation, and to make corrections for the evaluation of preoperative biometric indexes for reference.

ELIGIBILITY:
Inclusion Criteria:

(1) a diagnosis of myopia: equivalent spherical lens extent (SE) SE ≤ -0.0 D when the eye is relaxed in accommodation; (2) a diagnosis of cataract; (3) surgical treatment with sequential lens ultrasonoemulsification combined with monofocal IOL implantation in both eyes at our hospital; and (4) consent to participate and cooperate in this study.

Exclusion Criteria:

(1) Symptoms of acute eye diseases, such as eye redness, eye pain, and increased eye discharge; (2) Other binocular eye diseases that seriously affect visual function, such as amblyopia, glaucoma, diabetic retinopathy, severe age-related macular degeneration and retinal detachment; (3) Intra-operative or post-operative complications from cataract surgery; combined with other ophthalmologic surgeries; and any other ophthalmologic surgeries in both eyes during the follow-up period; (4) History of injuries; (5) Inability to understand the informed consent; and (6) Inability to communicate. ) history of trauma; (5) inability to understand the informed consent form and inability to communicate.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients (120 eyes) with high myopia who underwent binocular sequential lens ultrasonoemulsification combined with monofocal IOL implantation surgery for treatment of high myopia in our hospital were selected.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
pupil size | 1 week ,1 month, 3 months
  pupil size before and after surgery

IPD SHARING:
Plan to Share IPD: No